CLINICAL TRIAL: NCT01253109
Title: Detection of Induced IOP Fluctuations by SENSIMED Triggerfish® in Pigmentary Syndrome and Glaucoma Patients
Brief Title: Continuous Intraocular Pressure (IOP) Monitoring in Pigmentary Dispersion Syndrome and Pigmentary Glaucoma Patients
Status: Terminated | Type: Observational
Why Stopped: Law agreement between Triggerfish signal and GAT IOP during both sessions. However, an increase in the Triggerfish signal was observed during jogging phase.
Sponsor: Sensimed AG (Industry)
Collaborators: Private practicioner, Dr Sunaric Mégevand (Unknown); Orasis, AugenZentrum Pajic (Unknown)
Responsible Party: Jean-Marc Wismer, Sensimed AG
Other Study IDs: 09/11
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Pigmentary Dispersion Syndrome; Pigmentary Glaucoma Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SENSIMED Triggerfish
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Contact lens-based device for continuous IOP monitoring

SUMMARY:
This study monitors the intraocular pressure (IOP) over 4 to 6 hours using the SENSIMED Triggerfish® device and Goldmann Applanation Tonometry (GAT) in pigment dispersion syndrome and pigmentary glaucoma patients. The aim of the study is to detect SENSIMED Triggerfish® output signal peak after induced fluctuation by physical exercise or pupil dilation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pigmentary dispersion syndrome or pigmentary glaucoma on both eyes
* IOP of ≥ 15 mmHg
* 18-60 years.
* Patients able to jog continuously for at least 25 minutes
* Phakic eyes
* Patients who accept signing an informed consent approved by the Ethics Committee.

Exclusion Criteria:

* Pigmentary glaucoma already treated with peripheral laser iridotomy (PLI), argon laser peripheral iridoplasty (ALPI), argon laser trabeculoplasty (ALT) and selective laser trabeculoplasty (SLT) in any eye
* Patients treated with pilocarpine or other mydriatic agent within the last 4 weeks in any eye
* Anti-hypertensive treatment in the 4 weeks preceding the study and throughout the study. Following signature of informed consent, anti-hypertensive treatment will be washed out for 4 weeks prior to study procedures in enrolled patients
* Patients with pseudoexfoliative (PEX) syndrome or PEX glaucoma in any eye
* Patients not able to understand the nature of the research
* Patients under tutorship
* Corneal abnormality
* Subjects with contraindications for wearing contact lenses
* Full frame metal glasses during SENSIMED Triggerfish® monitoring
* History of other ocular surgery except uncomplicated strabismus surgery no later than 3 months prior to study procedures
* Ocular inflammation or infection
* History of cardiac or pulmonary disorder
* Pregnancy and lactation
* Simultaneous participation in other clinical research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with confirmed diagnosis of pigmentary dispersion syndrome or pigmentary glaucoma on both eyes
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
SENSIMED Triggerfish output values | during 4 to 6 hours
  Patients will undergo 2 sessions of 4 to 6 hours SENSIMED Triggerfish continuous intraocular pressure monitoring in a selected eye, during and/or after physical exercise and pupile dilation
Goldmann Applanation Tonometry values | During 4 to 6 hours
  GAT IOP readings will be done in the other eye at regular intervals during 4 to 6 hours SENSIMED Triggerfish IOP monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Sunaric Megevand, Dr, Principal Investigator — Private Practice
Locations (1):
- Private practice - Dr Sunaric Mégevand, Geneva, Switzerland